CLINICAL TRIAL: NCT06026345
Title: The Affera Global Registry is a Prospective, Global, Multi-center, Observational Post-market Registry (PMR)
Brief Title: Affera Global Registry
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: Affera Global Registry
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment Arm: Patients enrolled and treated with the Affera Platform
  Interventions: Device: Affera Platform

INTERVENTIONS:
Device: Affera Platform — A cardiac ablation will be performed using the Affera Platform

SUMMARY:
The Affera Global Registry is a prospective, global, multi-center, observational post-market registry (PMR). The purpose of this study is to describe clinical performance and safety data in a broad patient population treated with the Affera Platform.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age or minimum age as required by local regulations
* Planned procedure using the commercially available Affera Platform
* Willing and able to comply with study requirements and give IC (defined as legally effective, documented confirmation of a subject's voluntary agreement to participate in this clinical study) or authorization per institution and geographical requirements

Exclusion Criteria:

* Subject is enrolled in a concurrent study that has not been approved for concurrent enrollment by the global study manager
* Subject with exclusion criteria required by local law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years of age (or minimum age as required by local regulations) who have a recommendation for an ablation with the Affera Platform may be approached regarding enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective #1 (Efficacy) | 12 Month Post Proceedure
  Estimate freedom from recurrence of the arrhythmia(s) treated at the study index ablation procedure using the Affera Platform.

SECONDARY OUTCOMES:
Primary Objective #2 (Safety) | 90 Days Post Proceedure
  Estimate serious device and serious procedure-related adverse events for the Affera Platform.

CONTACTS AND LOCATIONS:
Locations (12):
- Universitair Ziekenhuis Brussel, Brussels, Belgium
- Czechia (2):
  - IKEM - Institut Klinické a Experimentální Medicíny, Prague
  - Nemocnice Na Homolce, Prague
- France (2):
  - Hôpital Haut-Lévêque - CHU de Bordeaux, Bordeaux
  - Clinique Pasteur, Toulouse
- Germany (3):
  - Charité Universitätsmedizin Berlin, DHZC - Campus Charité Mitte, Berlin
  - MVZ CCB Frankfurt und Main Taunus GbR, Frankfurt
  - Universitäres Herzzentrum, Hamburg
- Beacon Hospital, Dublin, Ireland
- Inselspital - Universitätsspital Bern, Bern, Switzerland
- United Kingdom (2):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No